CLINICAL TRIAL: NCT01978106
Title: Comparisons of the Astigmatic Power of Toric Intraocular Lens Using Three Toric Calculators: AcrySof, TECNIS, and iTrace Toric Calculator
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2013-0041
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Cataract; Astigmatism
Keywords: toric calculator; toric intraocular lens power; Acrysof; Tecnis; iTrace
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- a WTR corneal astigmatism group: Corneal astigmatism was defined as WTR when the steep corneal cylinder axis was within 30 degrees of the horizontal axis.
- an ATR corneal astigmatism group: Corneal astigmatism was defined as ATR when the cylinder axis was within 30 degrees of the vertical axis.

SUMMARY:
Purpose of this study is to compare the astigmatic power of the toric IOL obtained from the AcrySof toric calculator, TECNIS toric calculator, and iTrace toric calculator in a group of patients with preoperative with-the-rule (WTR) and against-the-rule (ATR) corneal astigmatism. The study included 100 eyes with cataract and greater than 0.75 diopter of corneal astigmatism, and the subjects were divided into WTR and ATR group. Keratometric value was measured using autokeratometry, IOLMaster partial coherence interferometry (PCI), iTrace incorporating corneal topography and ray-tracing aberrometry. Based on measured values, toric IOL power calculations were performed using AcrySof, TECNIS and iTrace toric calculators.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who planned to undergo cataract removal by phacoemulsification
* Subjects with preoperative corneal astigmatism greater than 0.75 D, as determined by autokeratometry

Exclusion Criteria:

* Subjects with more than 2.74 D of corneal keratometric value from autokeratometry
* a history of intraocular or corneal surgery and ocular trauma
* biomicroscopic evidence of corneal disease that could affect corneal astigmatisms
* contact lens wearer

Ages: 33 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who planned to undergo cataract removal by phacoemulsification between January 2013 to April 2013 at the Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea were included in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Difference of toric intraocular lens power between three toric calculators | Immediately after measurement
  Comparison of the toric intraocular lens power calculated from Acrysof and TECNIS toric calculators using keratometric values measured by autokeratometry or IOLMaster PCI and that from iTrace toric calculator with keratometric value measurement using iTrace ray tracing wavefront aberrometry and iTrace simulated keratometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea